CLINICAL TRIAL: NCT04853355
Title: Non-Responsive Diabetic Macular Edema in Patients With Pachychoroid and Choroidal Hyperpermeability.
Brief Title: Non-Responsive Diabetic Macular Edema and Spironolactone
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00073697
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Maculopathy
Keywords: spironolactone; anti-VEGF injections; aflibercept; Eylea
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spironolactone Treatment (Experimental): Patients with non-responsive Diabetic Macular Edema will be treated with Spironolactone in addition to the regular course of monthly aflibercept (Eylea).
  Interventions: Drug: Spironolactone 50 mg

INTERVENTIONS:
Drug: Spironolactone 50 mg — Add Spironolactone 50 mg to previous regimen

SUMMARY:
Diabetic patients with macular edema and choroidal hyperpermeability (as manifested as a thick choroid on OCT (optical coherence tomography) and ICG hyperfluorescence on ICG) unresponsive to anti-VEGF (vascular endothelial growth factor) and steroid injections will be treated with spironolactone in addition to the continued treatment of anti-VEGF injections, specifically aflibercept (Eylea).

DETAILED DESCRIPTION:
This is a non-randomized, prospective study of 10 patients referred during the years 2018 to 2020 with the diagnosis of Diabetic Macular Edema. Each patient was noted to have pachychoroid, choroidal hyperpermeability, and most important resistant to multiple anti-VEGF and steroid intravitreal injections, and have moderate vision loss. In addition, despite the fact that we use anti-VEGF medications, we do not know the levels of VEGF in the eye, nor do we have an explanation for the inability to respond to these drugs. This study will determine the degree of VEGF concentrations, response to anti-VEGF treatments, and determine biomarkers of inflammation as a means for explaining the cause of treatment resistance. Subsequently, another pathological process will be treated with spironolactone to see if the degree of contribution of choroidal hyperpermeability to the exudative process.

ELIGIBILITY:
Inclusion:

1. Presence of persistent Diabetic cystoid macular edema despite course of anti-VEGF injections and intraocular steroids. At the time of study baseline, the patients must be on q4 week intravitreal anti-VEGF medications and have failed (poor response - less than 50% decrease in macular central subfield thickness (CST) and volume) with intravitreal steroids (triamcinolone acetonide or dexamethasone implant).
2. Evidence of pachychoroid (choroid greater than 300 microns on OCT - EDI) with pachyvessels on OCT or OCTA. In addition, ICG (Indocyanine Green Angiogram) must show evidence of hyperfluorescence.
3. Visual Acuity of 20/25 to 20/400 at screening and baseline visits using an autorefractor or Early Treatment Diabetic Retinopathy Study (ETDRS).
4. IOP ≤ 25 mmHg - Patients that screen fail due to elevated IOP ˃25 mmHg may rescreen once IOP is treated and within normal limits (≤25 mmHg).

Exclusion:

1. Exudative maculopathies due to myopic choroidal degeneration, histoplasmosis, trauma, and specifically, the presence of angioid streaks.
2. Myocardial infarction or cerebrovascular accident within the last 6 weeks
3. Previous vitrectomy
4. Hypokalemia
5. Optic neuropathy
6. Traction maculopathies
7. Allergies to fluorescein and indocyanine, dilating agents, spironolactone, triamcinolone or anti-VEGF medications

   -

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of eyes with complete reabsorption of intraretinal fluid | 1 year
Macular Edema - Central Subgroup Thickening | 1 year
Macular Edema - Volume | 1 year
  Macular volume
Vision, best corrected, logMAR units | 1 year

SECONDARY OUTCOMES:
Extrafoveal exudation (nCST) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Nelson, MD MBA, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after completion date
Access Criteria: Contact Principal investigator

REFERENCES:
- [Background] Kim DY, Lee JY, Lee EK, Kim JY. COMPARISON OF VISUAL/ANATOMICAL OUTCOMES AND RECURRENCE RATE BETWEEN ORAL SPIRONOLACTONE AND PHOTODYNAMIC THERAPY FOR NONRESOLVING CENTRAL SEROUS CHORIORETINOPATHY. Retina. 2020 Jun;40(6):1191-1199. doi: 10.1097/IAE.0000000000002507. PMID 30897068